CLINICAL TRIAL: NCT05461859
Title: Right Anterior Ganglionated Plexus Ablation Without Pulmonary Vein Isolation for the Treatment of Vagally-mediated Paroxysmal Atrial Fibrillation.
Brief Title: Cardioneuroablation for the Treatment of Vagally-mediated Atrial Fibrillation.
Status: Completed | Type: Observational
Sponsor: St. Joseph's Centre, Poland (Other)
Responsible Party: Principal Investigator, Piotr Futyma, Associate Professor, St. Joseph's Centre, Poland
Other Study IDs: 42/2022/B
Record Dates: First submitted 2022-07-12; First posted 2022-07-18 (Actual); Last update posted 2023-11-27 (Actual); Status verified 2023-11

CONDITIONS: Atrial Fibrillation Paroxysmal
Keywords: Atrial Fibrillation; Vagally-mediated; Cardioneuroablation
MeSH Terms: conditions — Atrial Fibrillation | interventions — Calcineurin

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- ≥30% HR increase after CNA: Patients in whom ≥30% increase in HR after CNA of RAGP was achieved.
  Interventions: Procedure: Cardioneuroablation (CNA) of the right anterior ganglionated plexus (RAGP)
- <30% HR increase after CNA: Patients in whom ≥30% increase in HR after CNA of RAGP was *not* achieved.
  Interventions: Procedure: Cardioneuroablation (CNA) of the right anterior ganglionated plexus (RAGP)

INTERVENTIONS:
Procedure: Cardioneuroablation (CNA) of the right anterior ganglionated plexus (RAGP) — CNA of RAGP

SUMMARY:
Pulmonary vein isolation (PVI) is a cornerstone for catheter ablation of atrial fibrillation (AF), however, exact mechanisms of PVI efficacy remain debatable. It has been postulated that in patients with increased vagal tone AF can be treated by attenuation of parasympathetic drive to the heart using cardioneuroablation (CNA) by means of radiofrequency (RF) of the ganglionated plexi, however, data in literature and guidelines are lacking. The objective of this study is to examine the mid-term efficacy of RF-CNA targeting the right anterior ganglionated plexus (RAGP) in management of AF using right-atrial approach only.

DETAILED DESCRIPTION:
Calculation of deceleration capacity (DC) was derived from the result of 1-minute monitoring of R-R intervals recorded using electrophysiology (EP) system.

Double access to the right femoral vein was obtained under ultrasound guidance. Four- or ten-pole diagnostic electrode was introduced into the coronary sinus and an open-irrigated or 8 mm ablation catheter (AC) was advanced into the superior vena cava. The location of RAGP was determined purely anatomically at the sites of fragmented potentials below the superior vena cava ostium and the superior-septal aspect of the right atrium in the left anterior oblique (LAO) view and was guided fluoroscopically. RF applications were delivered and were continued until heart rate (HR) acceleration >30% was achieved or RF time exceeded 120 s.

Clinical follow-up (FU) consisted of multiple ambulatory visits with standard ECG and a 7-day Holter during the FU period. During FU visits, a detailed history of any palpitations, episodes of AF, and hospitalizations for cardiac arrhythmias was collected.

ELIGIBILITY:
Inclusion Criteria:

* Paroxysmal atrial fibrillation
* Deceleration capacity >7ms

Exclusion Criteria:

* Permanent AF lasting more than one year or persistent AF lasting more than 7 days
* AF secondary to electrolyte imbalance, thyroid disease, alcohol abuse, or other non-heart related causes
* Anteroposterior dimension of the left atrium in the echocardiography ≥ 5.5 cm
* Significant valvular disease
* Prosthetic valve
* Heart failure New York Heart Association (NYHA) class III/IV
* Previous AF ablation
* History of a persistent oval opening/atrial septal defect closure
* History of left atrial appendage closure
* Atrial myxoma
* Presence of a cardiac pacemaker, defibrillator or cardiac resynchronization therapy device
* Symptomatic hypotension
* History of pericarditis
* Congenital heart disease
* History of coagulation disorders
* Contraindications to oral anticoagulation
* Contraindications to computed tomography or magnetic resonance imaging
* History of transplantation
* Severe lung disease
* Chronic renal failure defined as estimated glomerular filtration rate (eGFR) <30 mL/min/m2
* Cancer
* Significant infection
* Life expectancy less than one year
* Lack of informed consent to participate in the trial
* Participation in another trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive patients with paroxysmal AF who were scheduled for ablation of AF and in whom clinical parameters such as sinus bradycardia and AF paroxysms occurring during rest, night or after meals, suggested vagally-mediated AF, were considered for the study.
Sampling Method: Probability Sample
Enrollment: 18 (Actual)
Dates: Start 2020-03-16 (Actual); Primary Completion 2021-07-19 (Actual); Study Completion 2023-01-01 (Actual)

PRIMARY OUTCOMES:
AF recurrence | 1 year
  AF episode lasting 30s or more, documented on 12-lead ECG, event or Holter monitor

CONTACTS AND LOCATIONS:
Locations (1):
- St. Joseph's Heart Rhythm Center, Rzeszów, Poland